CLINICAL TRIAL: NCT06499467
Title: Norepinephrine Equivalent Dose of Vasopressin, Phenylephrine and Epinephrine in Septic Shock Patients: A Prospective Study
Brief Title: Norepinephrine Equivalent Dose of Vasopressin, Phenylephrine and Epinephrine in Septic Shock
Status: Recruiting | Type: Observational
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Mohan Gurjar, Professor, Sanjay Gandhi Postgraduate Institute of Medical Sciences
Other Study IDs: 2024-112-DM-138
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Septic Shock
Keywords: Septic shock; Vasopressor Agent; Norepinephrine
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Septic shock is the most common form of circulatory shock encountered in patients admitted in intensive care unit. The initial management involves fluid resuscitation but if hypotension does not get resolved solely by it, then vasopressors become the mainstay of the management of shock to maintain adequate mean arterial pressure (MAP).

Norepinephrine is recommended as the first line vasopressor in the management of septic shock as per Surviving Sepsis Campaign guidelines of 2021. It recommends addition of vasopressin to the regime if the target MAP is not achieved with just norepinephrine. However, in clinical practice various other vasopressors are being used in the management of septic shock, as per clinical condition. Different vasopressors have different modes of action and pharmacological effects on hemodynamics. Therefore, there evolved the need of development of a formula that would reflect the potency of each vasopressor in a standardized manner. Thus, the concept of Norepinephrine Equivalence (NEE) came into existence. In the recent years, different studies were conducted in various parts of the world with different primary objectives. These authors have proposed different formulas for calculation Norepinephrine Equivalence (NEE) dose of the used vasopressors as an inference from their studies. All these formulas are based on assumptions and there lacks standardization. There are presently no studies available in the existing literature, where a prospective study is done to primarily determine the Norepinephrine equivalence dose (NEE) of other vasopressors in patients of septic shock. Hence, the investigators aim to find out equivalent dose of these different drugs, which are being used commonly in the management of septic shock, in a prospective planned study.

DETAILED DESCRIPTION:
Sepsis is a life-threatening state of organ dysfunction caused by dysregulated response of host to infection. It is the most common form of circulatory shock encountered in patients admitted in intensive care unit. In physiological state, blood pressure is maintained by the interplay of three major mechanisms namely sympathetic nervous system, vasopressin system and renin aldosterone system. However in the states of vasodilatory shock, these homeostatic mechanisms are disturbed. The initial management involves fluid resuscitation but if hypotension doesn't get resolved solely by it, then vasopressors become the mainstay of the management of shock to maintain adequate mean arterial pressure (MAP).

Norepinephrine has been recommended as the first line vasopressor for management of septic shock since 2004 and the latest guideline recommends addition of vasopressin along with norepinephrine when the target MAP is not achieved. However, in clinical practice various other vasopressors are used in the management of septic shock. Different vasopressors have different modes of action and pharmacological effects on hemodynamics. Therefore, there evolved the need of development of a formula that would reflect the potency of each vasopressor in a standardized manner. Thus, the concept of Norepinephrine Equivalence (NEE) came into existence. It is a scale to quantify the exposure to various vasopressors, by converting their dose as an equivalent of norepinephrine. It allows us to combine the dose of other vasopressors in a single scale and quantitatively assess the severity of shock when norepinephrine is being used along with other vasopressors.

Annane et al conducted a study in 2007 in 330 patients of septic shock with the primary objective of comparing the efficacy and safety of norepinephrine plus dobutamine with those of epinephrine alone in septic shock. They inferred from their study that the doses of vasopressors needed to achieve the MAP target were same for epinephrine and norepinephrine. Similarly, Myburgh et al studied in 280 patients of circulatory shock in the year 2008 to determine whether there was any difference between epinephrine and norepinephrine in achievement of MAP goal in the ICU patients and found that the maximal daily infusion of epinephrine and norepinephrine didn't have difference to achieve a target MAP. De Becker et al conducted a study in 2003 on 20 septic shock patients with the primary objective to assess the effects of different doses of dopamine, norepinephrine and epinephrine on the splanchnic circulation in patients of septic shock. They found that the final infusion rate of epinephrine was 0.62 mcg/kg/min, which was comparable to 0.45 mcg/kg/min rate of norepinephrine infusion to achieve the target MAP, suggesting a conversion ratio of 1.4:1. Hussain et al found in their study on 42 patients of septic shock in 2014 to determine the efficacy of phenylephrine in comparison to norepinephrine in patients of septic shock in ICU, that phenylephrine was 1.1 times equipotent to norepinephrine. Gordon et al studied on 409 patients of septic shock in 2016 to compare the effect of early vasopressin versus norepinephrine on kidney failure. They concluded from their study that 0.04U/min of vasopressin to be equivalent to 0.1 mcg/kg/min of norepinephrine.

Goradia et al proposed a norepinephrine equivalent formula in 2021 in their review article as Norepinephrine dose (mcg/kg/min) + epinephrine dose (mcg/kg/min) + 2.5 x vasopressin (U/min) + 0.1 × phenylephrine dose (mcg/kg/min). Kotani et al proposed a different norepinephrine equivalent formula in 2023 as follows Norepinephrine dose (µg/kg/min) + epinephrine dose (µg/kg/ min) + 0.06 × phenylephrine dose (µg/kg/min) + 2.5 × vasopressin dose (U/min).

However, since these calculations of NEE are based on assumptions and not standardized, there are several different formulae for calculation of the same. Different studies were conducted in different parts of the world with different primary objectives, the authors proposed different NEE formulas of the used vasopressor as an inference from their studies.

Presently, there are no studies available in the existing literature where a prospective study is done to primarily determine the Norepinephrine equivalence of other vasopressors namely vasopressin, phenylephrine and epinephrine, in patients of septic shock. Hence, the investigators aimed to study the NEE dose of the commonly used vasopressors in the ICU in septic shock patients.

During the study period, all adult ICU patients having septic shock will be considered for inclusion. Once the patient meets the inclusion/exclusion criteria, informed written consent will be obtained at the beginning of the study. The weight of the patient will be noted from the weight-measuring beds and the drug preparations are made accordingly. The transducer will be zeroed to the atmospheric pressure and baseline MAP will be recorded. A second vasopressor will be connected to the central venous catheter (CVC) as per the standard preparation. Then Norepinephrine infusion dose will be deescalated over 5-10 minutes by 0.1 mcg/kg/min. Simultaneously, the dose of the second vasopressor will be titrated to achieve the baseline MAP (±1 mmHg). Two readings of the dose of the second vasopressor will be recorded at least 5 minutes apart and their mean will be calculated. Evaluation with more than one vasopressor will depend upon the clinical condition of the patient as decided by the treating team. However, if more than one vasopressor are being assessed for NEE dose, then the next drug will be assessed after at least one hour gap. The same patient can be included for the study for more than once if they receive norepinephrine in three different dose ranges viz 0.1-0.5 mcg/kg/min, 0.5-1 mcg/kg/min and >1 mcg/kg/min.

Demographic and clinical characteristics of included patients will be recorded in structured case report forms. Candidates who qualify for the inclusion criteria will be included in the study. The baseline MAP will be recorded. The norepinephrine infusion will be tapered down gradually by 0.1 mcg/kg/min and in the meanwhile a second vasopressor will be introduced to maintain the baseline MAP recorded at the beginning of the study. After 15 minutes of stabilization of the dose of the second vasopressor, two readings of the dose of the second vasopressor will be taken 5 minutes apart and their mean will be taken as a NEE of that particular vasopressor.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients on mechanical ventilation in septic shock receiving norepinephrine in whom the treating clinical team plan to add another vasopressor, will be considered for inclusion if they meet these two condition (1) Patient is on Norepinephrine infusion at least 0.1 mcg/kg/min for the last 6 hours; and (2) There has been no dose alteration in the infusion of norepinephrine for the last 2 hours

Exclusion Criteria:

* There are concurrently other forms of shock like cardiogenic, obstructive, anaphylactic or hypovolemic.
* The patient has arrhythmias during the current course of illness.
* The patient has asynchrony on mechanical ventilator despite airway clearance with suctioning and adequate sedation at the time of study measurement.
* The patient is hypovolemic with ongoing fluid resuscitation in the form of fluid boluses, blood or blood product transfusions at the time of study measurement.
* The patient receives diuretic boluses or undergoes hemodialysis sessions at the time of study measurement.
* Pregnancy
* Patient who didn't consent for study or withdrew the consent at any point of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients on mechanical ventilation who are in septic shock condition receiving norepinephrine as vasopressor
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the norepinephrine equivalent dose of vasopressin, phenylephrine and epinephrine used in patients of septic shock. | Within 30 minutes of initiation of second vasopressor
  Norepinephrine will be gradually tapered by 0.1 mcg/kg/min over 10-15 minutes and simultaneously a second vasopressor will be introduced to maintain the baseline MAP (± 1 mm Hg). After stabilization for at least 5 minutes and achieving the same baseline MAP, two readings of the dose of the second vasopressor will be recorded, at least 5 min apart, and averaged. The averaged value of the second vasopressor dose will be considered as a NEE dose for that particular vasopressor against NE dose of 0.1 mcg/kg/min

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Gurjar, MD, PDCC, Principal Investigator — Sanjay Gandhi Postgraduate Institute of Medical Sciences (SGPGIMS)
Locations (1):
- Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: Undecided